CLINICAL TRIAL: NCT04546971
Title: Using Telehealth to Address Alcohol Misuse in HIV Care
Acronym: ReACH3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Christopher W. Kahler, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2P01AA019072 (NIH)
Record Dates: First submitted 2020-09-02; First posted 2020-09-14 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Drinking; HIV Viremia
MeSH Terms: conditions — Alcohol Drinking | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief intervention (Active Comparator): A brief alcohol intervention lasting about 10 minutes, delivered after the baseline assessments.
  Interventions: Behavioral: Brief Intervention
- Brief Intervention plus Telehealth Counseling (Experimental): A brief alcohol intervention followed by referral to a telehealth counseling protocol including 5 sessions of counseling based on Motivational Interviewing and delivered by videoconferencing. Telehealth counseling extends for up to two years and also includes a text messaging intervention to encourage reductions in drinking.
  Interventions: Behavioral: Brief Intervention; Behavioral: Telehealth Counseling; Behavioral: Text messaging

INTERVENTIONS:
Behavioral: Brief Intervention — Brief alcohol intervention delivered by telephone or videoconferencing focusing on advising participants to reduce drinking
Behavioral: Telehealth Counseling — 5 sessions of counseling on alcohol use based on Motivational Interviewing.
  Arms: Brief Intervention plus Telehealth Counseling
Behavioral: Text messaging — A daily and then monthly text messaging program designed to help participants monitor drinking, set goals, and reinforce successful reduction or abstinence.
  Arms: Brief Intervention plus Telehealth Counseling

SUMMARY:
This project will test the effects of a telehealth counseling program on reducing alcohol use and improving HIV viral control among people with HIV who drink heavily. In total, 600 heavy drinkers with HIV will be assigned to either (a) a single session of brief counseling on alcohol use or (b) brief counseling plus referral to a telehealth counseling program that includes multiple sessions of counseling by videoconferencing and text messaging support. To understand the effects of the program, participants' alcohol use, HIV outcomes, and health will be assessed over a 2-year period.

DETAILED DESCRIPTION:
The purpose of the proposed study is to test the real-world effectiveness of the ReACH (Reducing Alcohol use and related Comorbidities in HIV care) telehealth counseling protocol in a pragmatic Hybrid Type 1 effectiveness-implementation randomized trial. The study will recruit 600 heavy-drinking PLWH from four federally-qualified health centers in geographically distinct regions across the U.S, which provide services to over 14,000 PLWH. Upon completing enrollment, participants will be randomized to receive either single-session brief intervention (BI) by phone with referral to local treatment when appropriate or BI plus referral to ReACH telehealth counseling (TC). Participants will complete follow-ups through 24 months after baseline to assess longer-term changes in drinking and health outcomes. The study will test the hypothesis that TC compared to BI will result in (a) reduced number of drinks consumed per week and frequency of heavy drinking and (b) increased odds of having an undetectable viral load at 12- and 24-month follow-ups. Secondary outcomes include self-reported ART adherence, engagement in condomless sex with non-exclusive partners, frequency of other substance use, phosphatidylethanol levels (a biomarker of recent alcohol use), and Veterans Aging Cohort Study index scores. The study also will examine potential moderators of TC effectiveness. As a secondary aim, implementation measures corresponding to aspects of the Dynamic Sustainability Framework will be assessed including implementation outcomes of acceptability, appropriateness, and feasibility guided by Proctor's Implementation Outcomes Framework. Thus, this pragmatic Hybrid Type 1 trial will help establish the real-world effectiveness of the ReACH TC intervention while also providing key implementation-related measures and outcomes that will inform future ReACH TC scale up and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* In care for HIV at one of 4 participating federally qualified health centers, report at least one heavy drinking day (4+ drinks) or average more than 7 drinks per week in the past 30 days

Exclusion Criteria:

* need for supervised alcohol detoxification, as indicated by having a history of severe withdrawal symptoms such as seizures and delirium tremens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Alcoholics drinks consumed per week | 12 months
  Average number of alcoholic drinks consumed per week over the past 30 days
Alcoholics drinks consumed per week | 24 months
  Average number of alcoholic drinks consumed per week over the past 30 days
Number of heavy drinking days | 12 months
  Number of days consuming 4 or more drinks in a day over the past 30 days
Number of heavy drinking days | 24 months
  Number of days consuming 4 or more drinks in a day over the past 30 days
Proportion of participants with a detectable HIV viral load | 12 months
  Viral load test result that indicates HIV virus is detectable in the blood
Proportion of participants with a detectable HIV viral load | 24 months
  Viral load test result that indicates HIV virus is detectable in the blood

SECONDARY OUTCOMES:
Proportion of the past 30 days adherent to antiretroviral therapy | 12 months
  Antiretroviral therapy adherence as assessed by self-report
Proportion of the past 30 days adherent to antiretroviral therapy | 24 months
  Antiretroviral therapy adherence as assessed by self-report
Condomless sex with non-steady partners | 12 months
  Number of days in the past 30 having condomless sex with a non-steady partner
Condomless sex with non-steady partners | 24 months
  Number of days in the past 30 having condomless sex with a non-steady partner
Veterans Aging Cohort Study (VACS) index total score | 12 months
  Index of physiologic health calculated using HIV viral load, CD4 cell counts, liver function, creatinine, hemoglobin, platelets, white blood cell count, and height/weight (for body mass index). Higher scores indicate greater physiologic injury and risk for mortality.
Veterans Aging Cohort Study (VACS) index total score | 24 months
  Index of physiologic health calculated using HIV viral load, CD4 cell counts, liver function, creatinine, hemoglobin, platelets, white blood cell count, and height/weight (for body mass index). Higher scores indicate greater physiologic injury and risk for mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kahler, PhD, Principal Investigator — Brown University School of Public Health
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the National Data Archive. We also will post de-identified data used in the primary analyses of trial outcomes after those have been published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data in the NDA will be available 6 months after the first participants are recruited and will remain in there.
Access Criteria: Investigators can access date in the NDA using the available portal. We will allow access to the outcomes data to all through Brown's data archive once the outcome paper is published.